CLINICAL TRIAL: NCT03946150
Title: PaO2/FiO2*PEEP (P/FP) Ratio and Mortality in Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Sunitha PalaniDurai, Principal Investigator, National University Health System, Singapore
Other Study IDs: NUHSSingapore
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Adult Respiratory Distress Syndrome
Keywords: P/FP Ratio; ARDS Definition; Severity of Oxygenation in ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P/FP Ratio: P/FP Ratio is calculated in ARDS Patients retrospectively and analyse whether this new formula with PEEP can appropriately diagnose the Severity of Oxygenation with different levels of PEEP.
  Interventions: Diagnostic Test: P/FP Ratio
- P/F ratio: P/F ratio is the current Berlin definition of ARDS in Calculating the severity of Oxygenation.
  Interventions: Diagnostic Test: P/FP Ratio

INTERVENTIONS:
Diagnostic Test: P/FP Ratio — PaO2/Fio2 X PEEP

SUMMARY:
The PaO2/FiO2 (P/F) ratio is same for all the Positive End Expiratory Pressure (PEEP) ≥ to 5. This P/F ratio misleads the severity of disease without the knowledge of set PEEP. The Oxygenation status is actually worse when the patient is using high PEEP.

P/F Ratio doesn't include PEEP in the calculation.The P/F ratio doesn't show the severity of the disease appropriate for the set PEEP.

PaO2/(FiO2 X PEEP) P/FP Ratio is a new Formula which addresses this gap to appropriately calculate the severity of the disease by including PEEP in the formula.

This formula is used to predict mortality for different severities of ARDS.

DETAILED DESCRIPTION:
The Main aim of this study is to analyse whether this formula can early diagnose the severity of the disease appropriate for the set PEEP, so the Rescue measure can be started early which can eventually decreases the mortality.

Increasing the PEEP Value with the same Fio2 gives a different PaO2 and SpO2. The oxygenation improves substantially by increasing only the PEEP. So including the PEEP in calculating the severity of Oxygenation is better than the current practice.

The current Definition of ARDS for Oxygenation is P/F Ratio of 300 to 200 is Mild, 200 to 100 is Moderate and less than 100 is Severe ARDS with PEEP ≥ 5.

The New P/FP Ratio of 300 to 200 is mild, 200 to 100 is moderate and less than 100 is severe Adult Respiratory Distress Syndrome (ARDS) for all the different levels of PEEP values.

ELIGIBILITY:
Inclusion Criteria:

Intubated patients for

* Adult Respiratory Distress Syndrome
* Stroke
* Seizures
* Post neurosurgery
* Endoscopy Procedure
* Post Cardiac Collapse

Exclusion Criteria

Non intubated patients on

* Room Air
* Nasal Cannula
* Face mask
* Venturi Mask
* Non Rebreathing mask

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Intubated Patients admitted to ICU for ARDS and Non ARDS indications.
Sampling Method: Probability Sample
Enrollment: 4361 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
To predict mortality of ARDS patients using P/F and P/FP Ratio | Baseline ABG done at (approximately 4 hour after intubation) to ABG done approximately 1 hour before Rescue therapy like Neuro Muscular blockage, Proning, ExtraCorporeal Membrane Oxygenator, and High Frequency Oscillatory Ventilation.
  To predict mortality of different seventies of ARDS between P/F and P/FP Ratio. Day 1 ABG is taken and calulate the P/F and P/FP Ratio and analyze whether the new formula can predict the mortality on Day 1 after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha PalaniDurai, Principal Investigator — National University Health System, Singapore
Locations (1):
- National Universty Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palanidurai S, Phua J, Chan YH, Mukhopadhyay A. P/FP ratio: incorporation of PEEP into the PaO2/FiO2 ratio for prognostication and classification of acute respiratory distress syndrome. Ann Intensive Care. 2021 Aug 9;11(1):124. doi: 10.1186/s13613-021-00908-3. PMID 34370116